CLINICAL TRIAL: NCT06569459
Title: A Prospective, Randomized, Controlled, Single-center Phase II Clinical Trial of Trilaciclib Combined With Concurrent Chemoradiotherapy and Immunotherapy for Locally Advanced Esophageal Cancer.
Brief Title: Trilaciclib Combined With Concurrent Chemoradiotherapy and Immunotherapy in the Treatment of Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COSELA-ESCC-01
Record Dates: First submitted 2024-07-23; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — trilaciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Trilaciclib 240mg/m2；Radiation therapy：50.4Gy/28/1.8；Paclitaxel: 135mg/m2, d1, Q3W, 4 cycles；Carboplatin: AUC=5, d2, Q3W, 4 cycles（or nedaplatin 75 mg/m2, d2, Q3W, 4 cycles）;Immune inhibitors (by choice) : d1, Q3W, treatment + maintain phase, continuous dosing, until disease progression or not tolerated toxicity.
  Interventions: Drug: Trilaciclib Injection [Cosela]
- Control group (Sham Comparator): Radiation therapy：50.4Gy/28/1.8；Paclitaxel: 135mg/m2, d1, Q3W, 4 cycles；Carboplatin: AUC=5, d2, Q3W, 4 cycles（or nedaplatin 75 mg/m2, d2, Q3W, 4 cycles）;Immune inhibitors (by choice) : d1, Q3W, treatment + maintain phase, continuous dosing, until disease progression or not tolerated toxicity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trilaciclib Injection [Cosela] — Chemoradiotherapy and immunotherapy with Trilaciclib in the treatment of patients with unresectable locally advanced esophageal squamous cell carcinoma
  Other Names: G1T28; CDK 4/6 inhibitor
  Arms: Experimental group
Drug: Placebo — Chemoradiotherapy and immunotherapy in the treatment of patients with unresectable locally advanced esophageal squamous cell carcinoma
  Arms: Control group

SUMMARY:
This study is a double-arm, randomized, controlled, single-center, phase II clinical trial aimed at evaluating the efficacy and safety of chemoradiotherapy plus immunotherapy with or without Trilaciclib in the treatment of locally advanced esophageal squamous cell carcinoma that is not resectable.

DETAILED DESCRIPTION:
The subjects included in the study will receive Trilaciclib combined with chemoradiotherapy and immunosuppressant group ( the experimental group) and chemoradiotherapy combined with immunosuppressant group ( the control group). The experimental group and the control group were treated with 4 cycles of treatment. If the efficacy was evaluated as non-progressive after 4 cycles of treatment, the experimental group and the control group continued immunosuppressive therapy until disease progression or intolerance. The incidence of grade ≥3 neutropenia during chemotherapy was used as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participated in this study, signed the informed consent form, and had good compliance;
* Age ≥ 18 years old, male or female;
* Patients with histologically confirmed locally advanced esophageal squamous cell carcinoma at stage II-IV that is unresectable, or where surgery is contraindicated or refused (according to the AJCC 8th edition, the clinical stage before treatment was: cT1N2-3M0, cT2-4bN0-3M0, M1 limited to non-regional lymph node metastasis, excluding distant organ metastasis);
* The presence of at least one measurable lesion according to the response evaluation criteria in solid Tumors (RECIST1.1);
* Have not received any systemic anti-tumor therapy (including but not limited to systemic chemotherapy, radiotherapy, molecular targeted drug therapy, immunotherapy, biological therapy, local therapy, and other investigational therapeutic drugs);
* ECOG: 0-1 ;
* Expected survival time ≥ 6 months;
* Vital organ function meets the following requirements (no blood components and cell growth factors are allowed for 2 weeks before the start of screening examination) ：Absolute neutrophil count (ANC) ≥1.5×109/L；Platelet count ≥100×109/L；Hemoglobin ≥100 g/L in women or 110g/L in men；Serum albumin ≥2.8g/dL；Total bilirubin ≤1.5 × ULN and ALT, AST, and/or AKP≤2.5 × ULN

  , serum creatinine 1.5 x ULN or creatinine clearance or greater or less 60 ml/min (according to Cockcroft - Gault formula);
* International standardization ratio (INR) and part activated clotting time (APTT) live enzymes acuities were 1.5 x ULN (for the use of stable doses of anticoagulants such as: low molecular heparin or warfarin and INR within the scope of the expected treatment of anticoagulants can filter);
* Women: All women of childbearing potential must have a negative serum pregnancy test at screening and must be using reliable contraception from written informed consent until 3 months after last dose.

Exclusion Criteria:

* History of esophageal cancer surgery;
* Previous history of fistula caused by primary tumor invasion;
* High risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation;
* Subjects with poor nutritional status, who lost more than 10% of their body weight within 2 months before screening, had no significant improvement after nutritional intervention;
* major surgery or severe trauma within 4 weeks before the first dose of study drug;
* Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage; 7. Have received or are receiving any of the following：Anti-PD-1 or anti-PD-L1 antibody therapy, chemotherapy, radiotherapy, targeted therapy； received any study drug within 4 weeks before the first dose of the study drug； within 2 weeks before first use of the drugs need to be given corticosteroid (> 10 mg daily prednisone dose equivalent) or other immune inhibitors for treatment of the subjects system, except for local inflammation of the esophagus and prevent allergy and nausea, vomiting, use of corticosteroids；Have received an antitumor vaccine or a live vaccine within 4 weeks before the first dose of study drug;
* Have any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism); Patients with vitiligo or cured asthma/allergy in the same year era who did not need any intervention after adulthood were excluded. Patients with autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone and patients with type I diabetes treated with stable doses of insulin were eligible.
* A history of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation or allogeneic bone marrow transplantation;
* Subjects with uncontrolled cardiac clinical symptoms or diseases such as： (1) heart failure NYHA II or higher； (2) unstable angina ；(3) myocardial infarction within 1 year ；(4) clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
* Severe infection (CTC AE > 2) occurred within 4 weeks before the first dose of study drug, such as severe pneumonia requiring hospitalization, bacteremia, and infectious complications; Patients with active pulmonary inflammation on baseline chest imaging or signs and symptoms of infection requiring treatment with oral or intravenous antibiotics within 2 weeks before the first dose of study drug were excluded if prophylactic antibiotics were used.
* History of interstitial lung disease, non-infectious pneumonia, pulmonary function test confirmed ≥ grade 3 pulmonary dysfunction;
* Patients with active pulmonary tuberculosis infection detected by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or with a history of active pulmonary tuberculosis infection more than 1 year before enrollment but without regular treatment;
* The subject has active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive and HCV-RNA above the detection limit of the analytical method);
* There were more than grade 1 abnormal sodium, potassium, and calcium laboratory test values within 2 weeks before enrollment, which could not be improved after treatment;
* Allergy to any study drug or its components;
* Prior hematopoietic stem cell or bone marrow transplantation;
* Any other malignancy diagnosed before the first use of study drug, except those with a low risk of metastasis and death (5-year survival rate > 90%), such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ;
* Judging by the researchers, the participants have other factors that could lead to the forced midway termination of studies..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥3 neutropenia | during Trilaciclib plus chemotherapy assessed up to 84 days
  Incidence of grade ≥3 neutropenia

SECONDARY OUTCOMES:
Incidence of G-CSF treatment | during Trilaciclib plus chemotherapy assessed up to 1 years
  Incidence of G-CSF treatment
Incidence of platelet transfusion | during Trilaciclib plus chemotherapy assessed up to 1 years
  Incidence of platelet transfusion
Incidence of grade ≥3 anemia | during Trilaciclib plus chemotherapy assessed up to 84 days
  Incidence of grade ≥3 anemia
Incidence of grade ≥3 thrombocytopenia | during Trilaciclib plus chemotherapy assessed up to 84 days
  Incidence of grade ≥3 thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Ge, PHD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China